CLINICAL TRIAL: NCT04847895
Title: Observation of Treatment Patterns With Lucentis® (Ranibizumab) in Real-life Conditions in All Approved Indications
Brief Title: Observation of Treatment Patterns With Lucentis® in Real-life Conditions in All Approved Indications
Acronym: PACIFIC
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002ADE28
Record Dates: First submitted 2021-03-26; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration
Keywords: Lucentis; Ranibizumab; Neovascular (wet) age-related macular degeneration; nAMD; diabetic macular edema; retinal vein occlusions; choroidal neovascularizations
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lucentis: Patients administered Lucentis by prescription
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — There is no treatment allocation. Patients administered Lucentis by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This study is designed as an observational, non-interventional, multicenter, open label, single arm study in patients being treated with Lucentis® for any approved indication included in the local product posology.

DETAILED DESCRIPTION:
The prospective observation period per patient will be up to 24 months. A minimum of one follow-up visit per year is required in order to maintain patient's participation in the study.

The baseline visit will be used to assess eligibility and collect baseline characteristics information. The follow-up visits will take place at a frequency defined as per investigator's discretion.

The study eye is defined as the first eye treated during the study, the other eye will be considered as the fellow eye. If both eyes are treated at baseline, the right eye will be chosen as the study eye.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥18 years of age, being treated with Lucentis® for any approved indication in the local Lucentis® SmPC
* Written informed consent

Exclusion Criteria:

* As described in Lucentis® SmPC
* Participation in any other clinical study or NIS with Lucentis® as the investigational drug (such as OCEAN or LUMINOUS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients being treated with Lucentis® for any approved indication included in the local product posology. Patients will be enrolled from approximately 211 centers across Europe.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
mean change in visual acuity | Baseline, Up to month 24
  Visual acuity will be measured according to the method used by each participating physician in his/her routine practice. To be able to integrate different visual acuity assessment methods for analysis, visual acuity assessments performed using Snellen or decimal notation will be converted into an Early Treatment Diabetic Retinopathy Study (ETDRS) letter score equivalent.
mean change in central retinal thickness | Baseline, Up to month 24
  As central retinal thickness data is optional, this analysis will be performed only if data allow.

SECONDARY OUTCOMES:
Number of treatments | Up to 24 months
  Number of treatments will be provided
Number of visits | Up to 24 months
  Number of visits will be provided
Time interval between treatments | Up to 24 months
  Time interval between treatments will be provided
Time interval between visits | Up to 24 months
  Time interval between visits will be provided
Duration of treatment period | Up to 24 months
  Duration of treatment period will be provided
Maximum period of treatment extension | Up to 24 months
  Maximum period of treatment extension (where applicable)
Number of retreatments | Up to 24 months
  Number of retreatments will be provided
Reasons for retreatment | Up to 24 months
  Reasons for retreatment will be provided
Monitoring and treatment regimen - Therapy schemes | Up to 24 months
  The following therapy schemes are defined:
  * Fixed scheme (FIX): Planned interval of (control-) visits: "regular" and planned treatment performance: "at each visit"
  * Pro Re Nata (PRN): Planned interval of (control-) visits: "regular" and planned treatment performance: "as needed"
  * Treat & Extend (T+E): Planned interval of (control-) visits: "variable" and planned treatment performance: "at each visit"
  * Monitor & Extend (M+E): Planned interval of (control-) visits: "variable" and planned treatment performance: "as needed"
  FIX, PRN, T+E and M+E are based on documentation by visit regarding physician's planning and will be applied as overall planned therapy scheme, if no different therapy schemes are documented between patient's visit.
  Actual interval of (control-) visits and treatment performance will be derived using the documented visit dates and treatment documentations.
Reasons for choice of treatment regimen | Up to 24 months
  Reasons for choice of treatment regimen will be provided. The choice of treatment is described within 5 categories:
  * Medical reasons
  * Compability with organisation of practice/clinic
  * Compability with availability of patient
  * Patient's request
  * Other
Monitoring and treatment patterns as a function of health insurances | Up to 24 months
  The results from the above derived monitoring and treatment regimen will be stratified for German patients according to the status of insurance (public health insurance or private health insurance).
Number of treatments with Lucentis® vials and pre-filled syringe | Up to 24 months
  Number of treatments with Lucentis® vials and pre-filled syringe will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (135):
- Germany (120):
  - Novartis Investigative Site, Ettlingen, Baden-Wurttemberg
  - Novartis Investigative Site, Ahaus
  - Novartis Investigative Site, Andernach
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Arolsen-Meneringhausen
  - Novartis Investigative Site, Bad Liebenzell
  - Novartis Investigative Site, Bad Säckingen
  - Novartis Investigative Site, Baden-Baden
  - Novartis Investigative Site, Bautzen
  - Novartis Investigative Site, Beckum
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Borna
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Breisach
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Bremervörde
  - Novartis Investigative Site, Brühl
  - Novartis Investigative Site, Buchholz
  - Novartis Investigative Site, Buxtehude
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Cham
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Coswig
  - Novartis Investigative Site, Dannenberg
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eckental
  - Novartis Investigative Site, Ehingen
  - Novartis Investigative Site, Einbeck
  - Novartis Investigative Site, Erding
  - Novartis Investigative Site, Erkrath
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Frankenthal
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freudenstadt
  - Novartis Investigative Site, Friedberg
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Garching
  - Novartis Investigative Site, Glauchau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heppenheim an der Bergstrasse
  - Novartis Investigative Site, Herrsching am Ammersee
  - Novartis Investigative Site, Herzberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Hoppegarten
  - Novartis Investigative Site, Höhr-Grenzhausen
  - Novartis Investigative Site, Hösbach
  - Novartis Investigative Site, Jülich
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kempten
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Leer
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Meiben
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Mutterstadt
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neubrandenburg
  - Novartis Investigative Site, Neustadt
  - Novartis Investigative Site, Neustadt A. D. Weinstraße
  - Novartis Investigative Site, Neutraubling
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Obernkirchen
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Paderborn
  - Novartis Investigative Site, Peine
  - Novartis Investigative Site, Pfaffenhofen
  - Novartis Investigative Site, Pirna
  - Novartis Investigative Site, Plauen
  - Novartis Investigative Site, Polch
  - Novartis Investigative Site, Prien am Chiemsee
  - Novartis Investigative Site, Quakenbrück
  - Novartis Investigative Site, Raesfeld
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rhauderfehn
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Saarburg
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Salzgitter
  - Novartis Investigative Site, Schweinfurt
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sindelfingen
  - Novartis Investigative Site, Speyer
  - Novartis Investigative Site, Straubing
  - Novartis Investigative Site, Torgau
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Waldshut-Tiengen
  - Novartis Investigative Site, Wedel
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Wismar
  - Novartis Investigative Site, Worms
  - Novartis Investigative Site, Würzburg
- Netherlands (7):
  - Novartis Investigative Site, Bergen op Zoom, North Brabant
  - Novartis Investigative Site, Heerhugowaard, North Holland
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Terneuzen
  - Novartis Investigative Site, Tilburg
- Switzerland (8):
  - Novartis Investigative Site, Bern, Canton of Bern
  - Novartis Investigative Site, Neuchâtel, Canton of Neuchâtel
  - Novartis Investigative Site, Wil, Canton of St. Gallen
  - Novartis Investigative Site, Aarau
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: No